CLINICAL TRIAL: NCT02208492
Title: The Effects on Cognitive Function of Levetiracetam (Keppra®) Compared to Carbamazepine (Tegretol®, Carmazepine®) as Monotherapy for Children With Partial Seizure; A Multicentric Randomized Controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0365
Record Dates: First submitted 2014-08-03; First posted 2014-08-05 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Focal Epilepsy
Keywords: Levetiracetam, Carabamazepine
MeSH Terms: conditions — Epilepsies, Partial | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam (Experimental)
  Interventions: Drug: Levetiracetam
- Carabamazepine (Active Comparator)
  Interventions: Drug: Carabamazepine

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam is a second-generation antiepileptic drug that has been approved for the treatment of epilepsy in both children and adults. This anticonvulsant works by binding to the synaptic vesicle protein 2A resulting in a possible effect on neurotransmitter release from presynaptic vesicles, while the exact mechanism of action is still unclear. In both adults and children, levetiracetam treatment in has a proven efficacy in both localization-related and generalized epilepsies. In contrast to first generation, levetiracetam reports less side effects of somnolence or lethargy, but behavioral adverse events, such as changed mood state, aggression, and irritability are noted, but only a few studies have reported such effects in a systemic fashion.
  Arms: Levetiracetam
Drug: Carabamazepine — Carbamazepine, a first-generation antiepileptic medication, stabilizes the inactivated state of voltage-gated sodium channels, making fewer of these channels available to subsequently open, which leaves the affected cells less excitable and less seizure prone. It is approved for both focal seizures and generalized tonic-clonic or combined seizures for adults and children.
  Arms: Carabamazepine

SUMMARY:
Unlike the first generation antiepileptic medications, newer drugs for epilepsy such as levetiracetam are reported to have less adverse effect in children but not many studies have systematically reviewed the subject. This study aims to prospectively evaluate the effect of levetiracetam on neurocognition, behavioral issues and quality of life, as well as its seizure control efficacy and other adverse events in pediatric epilepsy patients, in comparison to carbamazepine, one of the classic antiepileptic medication, widely prescribed for both partial and generalized seizures, despite its well known side effects.

This multicenter, open-label, parallel-group trial is expected to enroll 130 patients from age 4 to 16 woh will be randomized into two groups, which will be prescribed with levetiracetam or carbamazepine. Series of neuropsychological assessment and behavioral and life evaluations of the patients will be performed at baseline period and after the 52 weeks of study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from age 4 to 16, who have been diagnosed with focal epilepsy
2. Patients who have experienced minimal two unprovoked seizures, or patients who have had one unprovoked seizure and have shown focal abnormality in the EEG
3. Patients who have not received any antiepileptic medications prior to the study (Those who have been treated with rescue medication are eligible)
4. Patients with eligible consent or with legal guardians have given official consent

Exclusion Criteria:

1. Patients with progressive CNS disease, or systemic illness
2. Patients with level of SGOT/SPGT above the doubled normal level or BUN/Creatinine above the 3 times of the normal range
3. Patients who had used other anti-epileptic medication during any period of the trial, including baseline period. (Benzodiazepine used as rescue therapy is acceptable)
4. Patients who show hypersensitive reaction to the study medication.
5. Patients with any psychological problems.
6. Patients deemed inappropriate for the study by the investigators

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Assessment and comparative analysis of initial and follow-up Neuropsychological evaluation in both treated groups. (Levetiracetam and Carbamazepine) | 52 weeks
  changes in a series of follow-up neurocognitive, behavioral, and emotional function tests (Korean Wechsler Intelligence Scale for Children-Third edition (K-WISC-III, for subjects 6-16 years old)19, 20 or the Korean Weschler Preschool and Primary Scale of Intelligence-Third edition (K-WIPSSI-III, for ages 4-6), Korean-Child Behavior Checklist (K-CBCL), Children's Depression Inventory (CDI) 24 and Revised Children's Manifest Anxiety Scale (RCMAS))

SECONDARY OUTCOMES:
Seizure control efficacy | 52 weeks
  Comparison of baseline frequency to final follow-up frequency during the last 24 weeks of the maintenance period(at last visit at 52 week time point)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Jung DE, Yu R, Yoon JR, Eun BL, Kwon SH, Lee YJ, Eun SH, Lee JS, Kim HD, Nam SO, Kim GH, Hwang SK, Eom S, Kang DR, Kang HC. Neuropsychological effects of levetiracetam and carbamazepine in children with focal epilepsy. Neurology. 2015 Jun 9;84(23):2312-9. doi: 10.1212/WNL.0000000000001661. Epub 2015 May 6. PMID 25948717